CLINICAL TRIAL: NCT03110848
Title: A Phase II, Open-labeled, Ophthalmological External Investigator-blinded, Single-center, Randomized, Superiority, Non Profit, Pilot Clinical Trial to Evaluate the Effects of Atorvastatin on Graves' Orbitopathy (GO) in Hypercholesterolemic Patients With Moderate-to-severe and Active GO Subjected to Intravenous Glucocorticoid Therapy: the STAGO Study
Brief Title: Effects of Atorvastatin in Graves' Orbitopathy (GO)
Acronym: STAGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Ricercatore (Assistant Professor), University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STAGO
Record Dates: First submitted 2017-03-23; First posted 2017-04-12 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Thyroid Associated Ophthalmopathy; Hypercholesterolemia
MeSH Terms: conditions — Graves Ophthalmopathy; Hypercholesterolemia | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Methylprednisolone

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Ophthalmologist blinded to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Statins (Experimental): Atorvastatin 20 mg daily associated with intravenous glucocorticoids, namely 500 mg of methylprednisolone weekly for 6 weeks, followed by 250 mg weekly for another 6 weeks, for a total dose of 4.5 mg.
  Interventions: Drug: Atorvastatin; Drug: Methylprednisolone
- No statins (Active Comparator): Intravenous glucocorticoids, namely 500 mg of methylprednisolone weekly for 6 weeks, followed by 250 mg weekly for another 6 weeks, for a total dose of 4.5 mg.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 20 mg daily
  Other Names: Statins
  Arms: Statins
Drug: Methylprednisolone — 500 mg of methylprednisolone weekly for 6 weeks, followed by 250 mg weekly for another 6 weeks, for a total dose of 4.5 mg.
  Other Names: Intravenous glucocorticoids

SUMMARY:
Graves' orbitopathy (GO) is the most common extra-thyroidal manifestation of Graves' disease (GD), being observed in ~25% of patients. Besides genetic and demographical variables, risk factors associated with the development of GO in GD patients are known to be inadequate control of hyperthyroidism, radioiodine treatment, and smoking. In a large retrospective study conducted in more than 8,000 individuals with GD it was observed that treatment with 3-hydroxy-3-methylglutaryl-coenzyme reductase inhibitors, better known as statins, is associated with a ~40% reduced risk of developing GO in GD patients. The findings were interpreted as the consequence of the anti-inflammatory action of statins, being GO notoriously an autoimmune, inflammatory conditions.

Statins are widely used for the treatment of hypercholesterolemia, for which they are quite effective. The possibility that their "protective" effect in terms of GO development in GD patients, as observed by Stein et al., was simply due to their hypolipemic actions was not considered. To evaluate the possibility that the findings reflected lowering of cholesterol rather than a direct anti-inflammatory effect of statins a prospective, observational study to assess the association between GO and high cholesterol levels and/or the relationship between the degree and/or activity of GO and hypercholesterolemia is ongoing. Preliminary findings suggest that GO is more severe and active in patients with high cholesterol levels. On the basis of these observations, the present randomized clinical trial was designed to be performed in hypercholesterolemic patients with GD and moderate-to-severe and active GO, aimed at investigating if lowering of cholesterol levels with statins is associated with a better outcome of GO.

ELIGIBILITY:
1. Informed consent
2. A diagnosis of Graves' disease
3. A moderately severe GO
4. Active GO
5. No corticosteroids or immunosuppressive treatment for GO in the last 3 months.
6. No previous surgical treatment for GO
7. No contraindication to GC
8. Male and female patients of age: 18-75 years
9. LDL-cholesterol levels of 115-189 mg/dl
10. No more than one cardiovascular risk factor (diabetes, high blood pressure, smoking, familial history of acute cardiovascular events, obesity)
11. Effective method of contraception
12. No mental illness that prevent patients from comprehensive, written informed consent
13. Compliant patient, regular follow-up possible

Exclusion Criteria:

1. lack of informed consent
2. Absence of Graves' hyperthyroidism (present or past)
3. Inactive GO
4. Optic neuropathy
5. Corticosteroids or immunosuppressive treatment for GO in the last 3 months.
6. Previous surgical treatment for GO
7. Contraindications to GC
8. Pregnancy, breast-feeding women
9. Acute or chronic liver disease
10. Hypersensitivity to atorvastatin or other statins, or hypersensitivity or intolerance to the medication excipients such as lactose.
11. Medications interfering/interacting with statins (CYP3A4 inhibitors or inductors)
12. Relevant Malignancy
13. Corticosteroids or other immunosuppressive agents within last 3 months
14. Recent (≤1 year) history of alcoholism or drug abuse
15. Clinical ASCVD (AthroSclerotic CardioVascular Disease)
16. LDL-cholesterol levels ≥190 mg/dl or presence of more than one associated cardiovascular risk factor (diabetes, high blood pressure, smoking, familial history of acute cardiovascular events, obesity)
17. Severe familial hyperlipemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Overall GO outcome determined using a composite evaluation | 6 months
  Overall GO outcome determined using a composite evaluation.
  A composite evaluation of GO was described previously.
  Possible outcomes are: improvement, worsening, no change, resulting in 3 categorical values
  Improvement: amelioration of two parameters in at least one eye, without deterioration of any parameters in both eyes:
  Deterioration: worsening in two parameters in at least one eye:
  All other cases are "no change"
  Parameters are:
  Eyelid swelling (improvement/worsening according to EUGOGO Atlas evaluation) Lid aperture in mm (significant variation: 2 or more mm) Clinical activity score (CAS) (7 items: spontaneous pain, evoked pain, eyelid edema, eyelid redness, conjunctiva redness, caruncle edema, chemosis; significant change: at least 2 points) Exophthalmos in mm (significant variation 2 or more mm) Eye muscle involvement - diplopia score (Gorman score) (significant variation: disappearance or change in the degree, or improvement of ≥12 degrees in motility)

SECONDARY OUTCOMES:
Overall GO outcome determined using a composite evaluation | 3 months
  Overall GO outcome determined using a composite evaluation.
  A composite evaluation of GO was described previously.
  Possible outcomes are: improvement, worsening, no change, resulting in 3 categorical values
  Improvement: amelioration of two parameters in at least one eye, without deterioration of any parameters in both eyes:
  Deterioration: worsening in two parameters in at least one eye:
  All other cases are "no change"
  Parameters are:
  Eyelid swelling (improvement/worsening according to EUGOGO Atlas evaluation) Lid aperture in mm (significant variation: 2 or more mm) Clinical activity score (CAS) (7 items: spontaneous pain, evoked pain, eyelid edema, eyelid redness, conjunctiva redness, caruncle edema, chemosis; significant change: at least 2 points) Exophthalmos in mm (significant variation 2 or more mm) Eye muscle involvement - diplopia score (Gorman score) (significant variation: disappearance or change in the degree, or improvement of ≥12 degrees in motility)
Comparison of a disease specific quality of life questionnaire (GO-QoL) | 6 months
  A GO-specific quality of life questionnaire (GO-QoL) comprises 16 items, 8 concerning appearance and 8 concerning function. The combination of the various parameters gives a final numeric value which will be compared between the two groups
Comparison of a disease specific quality of life questionnaire (GO-QoL) | 3 months
  A GO-specific quality of life questionnaire (GO-QoL) comprises 16 items, 8 concerning appearance and 8 concerning function. The combination of the various parameters gives a final numeric value which will be compared between the two groups
GO relapse | 6 months
  Worsening in comparison with the 3-month evaluation
Requirement for additional treatments | 3 months
  Additional intravenous glucocorticoids, radiotherapy, orbital decompression, immunosuppressive treatments of any kind
Requirement for additional treatments | 6 months
  Additional intravenous glucocorticoids, radiotherapy, orbital decompression, immunosuppressive treatments of any kind

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Cisanello-Endocrinology I and II, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lanzolla G, Sabini E, Leo M, Menconi F, Rocchi R, Sframeli A, Piaggi P, Nardi M, Marcocci C, Marino M. Statins for Graves' orbitopathy (STAGO): a phase 2, open-label, adaptive, single centre, randomised clinical trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):733-742. doi: 10.1016/S2213-8587(21)00238-2. Epub 2021 Sep 27. PMID 34592164